CLINICAL TRIAL: NCT00699114
Title: Analgesic Effect of Ibuprofen 400, 600 and 800 mg, Paracetamol 500 and 1000 mg, and Paracetamol 1000 mg Plus 60 mg Codeine: Single-dose, Randomized, Placebo-controlled and Double-blind Study on Acute Pain After Third Molar Surgery
Brief Title: Analgesic Effect of Ibuprofen, Paracetamol (Acetaminophen), and Paracetamol (Acetaminophen) Plus Codeine on Acute Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Professor Lasse A. Skoglund, DDS, DSci, University of Oslo
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARIBU-020
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Surgery
Keywords: Pain; Analgesics; Molar; Third; Acetaminophen; Paracetamol; Ibuprofen; Codeine; Placebo
MeSH Terms: conditions — Pain | interventions — Lactose; Ibuprofen; Acetaminophen; Codeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator): Single dose placebo capsule
  Interventions: Drug: Placebo
- Ibuprofen 400 mg (Active Comparator): Single dose ibuprofen 400 mg capsule
  Interventions: Drug: Ibuprofen 400 mg
- Ibuprofen 600 mg (Active Comparator): Single dose ibuprofen 600 mg capsule
  Interventions: Drug: Ibuprofen 600 mg
- Ibuprofen 800 mg (Active Comparator): Single dose ibuprofen 800 mg capsule
  Interventions: Drug: Ibuprofen 800 mg
- Paracetamol 500 mg (Active Comparator): Paracetamol 500 mg (acetaminophen) capsule
  Interventions: Drug: Paracetamol (acetaminophen) 500 mg
- Paracetamol 1000 mg (Active Comparator): Single dose paracetamol 1000 mg (acetaminophen) capsule
  Interventions: Drug: Paracetamol (acetaminophen) 1000 mg
- Paracetamol 1000 mg + codeine 60 mg (Active Comparator): Single dose paracetamol (acetaminophen) 1000 mg + codeine 60 mg capsule
  Interventions: Drug: Paracetamol (acetaminophen) 1000 mg + codeine 60 mg

INTERVENTIONS:
Drug: Placebo — Lactose as powder in gelatine capsules, single dose
  Other Names: Lactose
  Arms: Placebo
Drug: Ibuprofen 400 mg — Ibuprofen 400 mg as powder in gelatine capsules, single dose
  Other Names: M01A E01 Ibuprofen
  Arms: Ibuprofen 400 mg
Drug: Ibuprofen 600 mg — Ibuprofen 600 mg as powder in gelatine capsules, single dose
  Other Names: M01A E01 Ibuprofen
  Arms: Ibuprofen 600 mg
Drug: Ibuprofen 800 mg — Ibuprofen 800 mg as powder in gelatine capsules, single dose
  Other Names: M01A E01 Ibuprofen
  Arms: Ibuprofen 800 mg
Drug: Paracetamol (acetaminophen) 500 mg — Paracetamol (acetaminophen) 500 mg as powder in gelatine capsules, single dose
  Other Names: N02B E01 Paracetamol (acetaminophen)
  Arms: Paracetamol 500 mg
Drug: Paracetamol (acetaminophen) 1000 mg — Paracetamol (acetaminophen) 1000 mg as powder in gelatine capsules, single dose
  Other Names: N02B E01 Paracetamol (acetaminophen)
  Arms: Paracetamol 1000 mg
Drug: Paracetamol (acetaminophen) 1000 mg + codeine 60 mg — Paracetamol (acetaminophen) 1000 mg + codeine 60 mg as powder in gelatine capsules, single dose
  Other Names: N02B E01 Paracetamol (acetaminophen) + R05D A04 codeine
  Arms: Paracetamol 1000 mg + codeine 60 mg

SUMMARY:
The purpose of this placebo controlled clinical trial is to evaluate the dose response relationship of ibuprofen in doses from 400 mg to 800 mg and paracetamol (acetaminophen)in doses from 500 mg to 1000 mg compared with paracetamol (acetaminophen)1000 mg plus codeine 60 mg on acute postoperative pain after surgical removal of impacted third molars.

DETAILED DESCRIPTION:
Acetaminophen (paracetamol) and related aspirin-like drugs have traditionally been used for pain control of minor to moderate postoperative pain. Gradually traditional non-steroidal anti-inflammatory drugs (NSAIDs) have become more popular as analgesics due to assumed superior therapeutic effects and aggressive marketing campaigns orchestrated by the pharmaceutical industry.

Ibuprofen is a widely used analgesic both in non-prescription and prescription doses.

A dose-response relationship for low ibuprofen doses is shown. Evidence of a progressing dose response relationship for moderate (i.e. 400 mg) to higher doses is scarce. A possible analgesic ceiling effect has been suggested for doses above 400 mg, although a correlation between given ibuprofen doses above 400 mg and patient serum levels is shown. However, it may be questioned if the plasma concentration of ibuprofen is an important determinator of analgesic drug efficacy. A higher dose is more likely to influence the duration of analgesic effect rather than the peak analgesic effect.

There are few clinical trials investigating the dose-response relationship of increasing ibuprofen doses and paracetamol doses. To our knowledge no published study has investigated the dose-response relationship of ibuprofen and paracetamol in the same trial with a negative (i.e. placebo) and a positive (i.e. best standard analgesic treatment) control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes referred for surgical removal of impacted third molars, due to symptoms or after being advised to do so by their dentist.
* Persons of both sexes (ASA type I).
* Females who are not pregnant or plan conception.
* Persons who have not used analgesics for 3 days prior to the day of surgery.
* Persons without known active ulcus or gastrointestinal bleeding.
* Persons without any known hypersensitivity for NSAIDs.
* Persons under no other continuous drug treatment than contraceptives.
* Caucasian origin.
* Persons with at least moderate postoperative pain as defined by subjective score on a verbal rating scale after surgical removal of third molars.

Exclusion Criteria:

* Patients with surgery time exceeding 60 minutes
* Peroperative complications such as profuse bleeding or perforation to the maxillary sinus requiring additional drug treatment during or after the surgical removal of the third molar.
* Postoperative complications such as extended bleeding, nausea and regurgitation during the observation period.
* Smoking before taking the test-drug or during the observation period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sum Pain Intensity Score(SPI) | 3 hour observation period

SECONDARY OUTCOMES:
Sum Pain Intensity Difference Score (SPID) | 3 hours
Sum Pain Intensity Score (SPI) | 6 hours
Sum Pain Intensity Difference Score (SPID) | 6 hours
Maximum Pain Intensity Difference Score (MAXPID) | Unknown, calculated variable
Time to Maximum Pain Intensity Difference Score | Unknown, calculated variable
Self-reported Occurrence of Adverse Effects | 3 hours
Self-reported Occurrence of Adverse Effects | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lasse A Skoglund, DDS, DSCi, Study Chair — Section of Dental Pharmacology and Pharmacotherapy, ICD, Faculty of Dentistry, University of Oslo, POB 1119 Blindern, N-0317 Oslo, Norway; Per Skjelbred, MD, DDS, PhD, Study Director — Department of Oral and Maxillofacial Surgery, Ullevaal University Hospital, Kirkeveien 166, N-0407 Oslo, Norway; Gaute Lyngstad, DDS, Principal Investigator — Section of Dental Pharmacology and Pharmacotherapy, ICD, Faculty of Dentistry, University of Oslo, POB 1119 Blindern, N0317 Oslo, Norway
Locations (1):
- Department of Oral and Maxillofacial Surgery, Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Lyngstad G, Skjelbred P, Swanson DM, Skoglund LA. Analgesic effect of oral ibuprofen 400, 600, and 800 mg; paracetamol 500 and 1000 mg; and paracetamol 1000 mg plus 60 mg codeine in acute postoperative pain: a single-dose, randomized, placebo-controlled, and double-blind study. Eur J Clin Pharmacol. 2021 Dec;77(12):1843-1852. doi: 10.1007/s00228-021-03231-9. Epub 2021 Oct 16. PMID 34655316